CLINICAL TRIAL: NCT04964427
Title: The Effects of Methylphenidate (MPH) and Non-invasive Brain Stimulation (tDCS) on Inhibitory Control Children With Attention-Deficit/Hyperactivity Disorder (ADHD)
Brief Title: The Effects of Methylphenidate and Non-invasive Brain Stimulation on Inhibitory Control in Children With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Deny Menghini, Principal Investigator, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2185_2020_OPBG
Record Dates: First submitted 2021-07-01; First posted 2021-07-16 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: methylphenidate; executive functions; working memory; tDCS; inhibitory control
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Study participants will receive the three conditions in random order:
  * a single dose of immediate release MPH (Ritalin®) administered according to the AIFA and NICE guidelines for ADHD;
  * a single 1 mA anodal tDCS session over the DLPFC for 20 min
  * a single session of sham tDCS over the DLPFC for 30s at the beginning and end of the tDCS session.
  The order of administration of the conditions will be counterbalanced between the participants and the conditions will be spaced apart from an interval of 24 hours.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- anodal tDCS- sham tDCS- MPH (Experimental): (A) anodal tDCS at t1 (B) sham tDCS at t2 (C) MPH at t3
  Interventions: Drug: Methylphenidate; Device: anodal tDCS; Device: sham tDCS
- anodal tDCS- MPH- sham tDCS (Experimental): (A) anodal tDCS at t1 (C) MPH at t2 (B) sham tDCS at t3
  Interventions: Drug: Methylphenidate; Device: anodal tDCS; Device: sham tDCS
- sham tDCS- anodal tDCS- MPH (Experimental): (B) sham tDCS at t1 (A) anodal tDCS at t2 (C) MPH at t3
  Interventions: Drug: Methylphenidate; Device: anodal tDCS; Device: sham tDCS
- sham tDCS- MPH- anodal tDCS (Experimental): (B) sham tDCS at t1 (C) MPH at t2 (A) anodal tDCS at t3
  Interventions: Drug: Methylphenidate; Device: anodal tDCS; Device: sham tDCS
- MPH- anodal tDCS- sham tDCS (Experimental): (C) MPH at t1 (A) anodal tDCS at t2 (B) sham tDCS at t3
  Interventions: Drug: Methylphenidate; Device: anodal tDCS; Device: sham tDCS
- MPH- sham tDCS- anodal tDCS (Experimental): (C) MPH at t1 (B) sham tDCS at t2 (A) anodal tDCS at t3
  Interventions: Drug: Methylphenidate; Device: anodal tDCS; Device: sham tDCS

INTERVENTIONS:
Drug: Methylphenidate — A single dose of 5-10 mg of immediate release MPH (Ritalin®) will be administered in line with NICE and AIFA (Agenzia Italiana del Farmaco) guidelines for ADHD treatment.
  Other Names: Ritalin
Device: anodal tDCS — Anodal electrode will be positioned over the left dlPFC, according to the 10-20 EEG on the sites corresponding F3, whereas the reference electrode will be placed above the contralateral supraorbital area, corresponding to Fp2. In the active tDCS condition, the current will increase slowly during the first 30 seconds to 1 mA (ramp-up) and, at the end of the stimulation, the current will decrease slowly to 0 mA during the last 30 seconds (ramp-down). Between the ramp-up and ramp-down constant current will be delivered for 20 minutes, with a density of 0.04 mA/cm2.
Device: sham tDCS — In the sham tDCS condition, the stimulation will be delivered by using the same active tDCS montage, respectively left-anodal dlPFC and right-reference electrode over Fp2. Stimulation intensity will be set at 1 mA, but the current will be applied for 30 seconds and will be ramped down without the participants' awareness.

SUMMARY:
The aim of this study is comparing the effects of non-pharmacological intervention (transcranial Direct Current Stimulation, tDCS) with those of drug (methylphenidate, MPH) administration in children and adolescents with ADHD.

The investigators hypothesized that tDCS would improve inhibitory control and visuo-spatial working memory as well as MPH.

DETAILED DESCRIPTION:
A sham controlled within-subjects study design will be conducted. Clinical eligibility screening will be completed at baseline. All participants will undergo an extensive neuropsychiatric evaluation in which developmental neuropsychiatrists and psychologists will evaluate the cognitive and the adaptive level, the severity of ADHD symptoms, and the presence of comorbid psychiatric disorders. After completing baseline assessment (T0), participants will be exposure to 3 conditions with an intersession-interval of 24h (T1, T2, T3): A) a single administration of 1 milliampere (mA) anodal tDCS session over the dorsolateral prefrontal cortex (DLPFC); B) a single administration of 1 mA sham tDCS session over the DLPFC; C) a single administration of immediate release MPH (Ritalin®), in accordance with the National Institute for Clinical Excellence (NICE) guidelines for ADHD (NICE, 2000). The order of the conditions will be counterbalanced across participants. After recruitment, the participants will be assigned to one of the 6 possible combinations of conditions (ABC, ACB, BAC, BCA, CBA, or CAB). The assignment will be according to a randomization order generated by a computer. The randomization information will be maintained by an independent researcher until data collection is completed. Participants will be tested on inhibitory control, by the Stop Signal Task (SST) and on working memory, by the N-Back Task, at baseline (T0), during tDCS administration (after 10 minutes of anodal and sham conditions) and after 1 hour of MPH administration. To verify that carry-over effects will not occur, the SST and the N-Back Task will be performed before each session (T1, T2, T3) and results will be compared with those obtained at baseline (T0). If the participant will not return to baseline level, another evaluation will be administered at least after two hours and, again, until participant's performance will return to baseline. Participants and parents will be blinded to tDCS conditions allocation. The tDCS will be carried out with a BrainStim stimulator.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* Patients must receive a Diagnostic and Statistical Manual of Mental Disorders (DSM-5) oriented diagnosis of ADHD and need drug treatment for the severity of symptoms;
* Intelligent Quotient (IQ) > 85;

Exclusion Criteria:

* Presence of Autism Spectrum Disorders;
* Presence of Mood Disorders;
* Previous/current diagnosis of neurological conditions (i.e. epilepsy, neurodegenerative diseases);
* Presence of Genetic Syndromes;
* Presence of basal medical conditions (i.e. heart, kidney or liver diseases) which may exclude the possibility to administer MPH.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-10-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
evaluate the change in response inhibition measures | immediately after the interventions
  Compare Stop Signal Reaction Times in patients with ADHD following the administration of a single anodal tDCS session, a single sham tDCS session and a single dose of MPH

SECONDARY OUTCOMES:
evaluate the change in other response inhibition measures | immediately after the interventions
  Reaction Times and Variability of Reaction Times of SST in patients with ADHD following the administration of a single anodal tDCS session, a single sham tDCS session and a single dose of MPH
evaluate the change in visuo-spatial working memory measure | immediately after the interventions
  Compare N-Back Correct Scores of visuo-spatial working memory task in patients with ADHD following the administration of a single anodal tDCS session, a single sham tDCS session and a single dose of MPH

CONTACTS AND LOCATIONS:
Locations (1):
- Bambino Gesù Hospital and Research Institute, Roma, Italy

REFERENCES:
- [Result] Adamo N, Hodsoll J, Asherson P, Buitelaar JK, Kuntsi J. Ex-Gaussian, Frequency and Reward Analyses Reveal Specificity of Reaction Time Fluctuations to ADHD and Not Autism Traits. J Abnorm Child Psychol. 2019 Mar;47(3):557-567. doi: 10.1007/s10802-018-0457-z. PMID 30027330
- [Result] Adams ZW, Roberts WM, Milich R, Fillmore MT. Does response variability predict distractibility among adults with attention-deficit/hyperactivity disorder? Psychol Assess. 2011 Jun;23(2):427-36. doi: 10.1037/a0022112. PMID 21443365
- [Result] Andreou P, Neale BM, Chen W, Christiansen H, Gabriels I, Heise A, Meidad S, Muller UC, Uebel H, Banaschewski T, Manor I, Oades R, Roeyers H, Rothenberger A, Sham P, Steinhausen HC, Asherson P, Kuntsi J. Reaction time performance in ADHD: improvement under fast-incentive condition and familial effects. Psychol Med. 2007 Dec;37(12):1703-15. doi: 10.1017/S0033291707000815. Epub 2007 May 31. PMID 17537284
- [Result] Aron AR, Dowson JH, Sahakian BJ, Robbins TW. Methylphenidate improves response inhibition in adults with attention-deficit/hyperactivity disorder. Biol Psychiatry. 2003 Dec 15;54(12):1465-8. doi: 10.1016/s0006-3223(03)00609-7. PMID 14675812
- [Result] Arul-Anandam AP, Loo C, Sachdev P. Transcranial direct current stimulation - what is the evidence for its efficacy and safety? F1000 Med Rep. 2009 Jul 27;1:58. doi: 10.3410/M1-58. PMID 20948722
- [Result] Banaschewski T, Coghill D, Santosh P, Zuddas A, Asherson P, Buitelaar J, Danckaerts M, Dopfner M, Faraone SV, Rothenberger A, Sergeant J, Steinhausen HC, Sonuga-Barke EJ, Taylor E. Long-acting medications for the hyperkinetic disorders. A systematic review and European treatment guideline. Eur Child Adolesc Psychiatry. 2006 Dec;15(8):476-95. doi: 10.1007/s00787-006-0549-0. Epub 2006 May 5. PMID 16680409
- [Result] Barkley RA, Fischer M, Smallish L, Fletcher K. Young adult outcome of hyperactive children: adaptive functioning in major life activities. J Am Acad Child Adolesc Psychiatry. 2006 Feb;45(2):192-202. doi: 10.1097/01.chi.0000189134.97436.e2. PMID 16429090
- [Result] Bedard AC, Martinussen R, Ickowicz A, Tannock R. Methylphenidate improves visual-spatial memory in children with attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2004 Mar;43(3):260-8. doi: 10.1097/00004583-200403000-00006. PMID 15076258
- [Result] Bellgrove MA, Hester R, Garavan H. The functional neuroanatomical correlates of response variability: evidence from a response inhibition task. Neuropsychologia. 2004;42(14):1910-6. doi: 10.1016/j.neuropsychologia.2004.05.007. PMID 15381021
- [Result] Biederman J, Spencer T. Attention-deficit/hyperactivity disorder (ADHD) as a noradrenergic disorder. Biol Psychiatry. 1999 Nov 1;46(9):1234-42. doi: 10.1016/s0006-3223(99)00192-4. PMID 10560028
- [Result] BINDMAN LJ, LIPPOLD OC, REDFEARN JW. THE ACTION OF BRIEF POLARIZING CURRENTS ON THE CEREBRAL CORTEX OF THE RAT (1) DURING CURRENT FLOW AND (2) IN THE PRODUCTION OF LONG-LASTING AFTER-EFFECTS. J Physiol. 1964 Aug;172(3):369-82. doi: 10.1113/jphysiol.1964.sp007425. No abstract available. PMID 14199369
- [Result] Boggio PS, Ferrucci R, Mameli F, Martins D, Martins O, Vergari M, Tadini L, Scarpini E, Fregni F, Priori A. Prolonged visual memory enhancement after direct current stimulation in Alzheimer's disease. Brain Stimul. 2012 Jul;5(3):223-230. doi: 10.1016/j.brs.2011.06.006. Epub 2011 Jul 27. PMID 21840288
- [Result] Boonstra AM, Kooij JJ, Oosterlaan J, Sergeant JA, Buitelaar JK. Does methylphenidate improve inhibition and other cognitive abilities in adults with childhood-onset ADHD? J Clin Exp Neuropsychol. 2005 Apr;27(3):278-98. doi: 10.1080/13803390490515757. PMID 15969353
- [Result] Brunoni AR, Amadera J, Berbel B, Volz MS, Rizzerio BG, Fregni F. A systematic review on reporting and assessment of adverse effects associated with transcranial direct current stimulation. Int J Neuropsychopharmacol. 2011 Sep;14(8):1133-45. doi: 10.1017/S1461145710001690. Epub 2011 Feb 15. PMID 21320389
- [Result] Buzy WM, Medoff DR, Schweitzer JB. Intra-individual variability among children with ADHD on a working memory task: an ex-Gaussian approach. Child Neuropsychol. 2009 Sep;15(5):441-59. doi: 10.1080/09297040802646991. PMID 19184779
- [Result] Cachoeira CT, Leffa DT, Mittelstadt SD, Mendes LST, Brunoni AR, Pinto JV, Blazius V, Machado V, Bau CHD, Rohde LA, Grevet EH, Schestatsky P. Positive effects of transcranial direct current stimulation in adult patients with attention-deficit/hyperactivity disorder - A pilot randomized controlled study. Psychiatry Res. 2017 Jan;247:28-32. doi: 10.1016/j.psychres.2016.11.009. Epub 2016 Nov 10. PMID 27863315
- [Result] Castellanos FX, Sonuga-Barke EJ, Scheres A, Di Martino A, Hyde C, Walters JR. Varieties of attention-deficit/hyperactivity disorder-related intra-individual variability. Biol Psychiatry. 2005 Jun 1;57(11):1416-23. doi: 10.1016/j.biopsych.2004.12.005. Epub 2005 Jan 28. PMID 15950016
- [Result] Castells X, Ramos-Quiroga JA, Rigau D, Bosch R, Nogueira M, Vidal X, Casas M. Efficacy of methylphenidate for adults with attention-deficit hyperactivity disorder: a meta-regression analysis. CNS Drugs. 2011 Feb;25(2):157-69. doi: 10.2165/11539440-000000000-00000. PMID 21254791
- [Result] Chabot RJ, Orgill AA, Crawford G, Harris MJ, Serfontein G. Behavioral and electrophysiologic predictors of treatment response to stimulants in children with attention disorders. J Child Neurol. 1999 Jun;14(6):343-51. doi: 10.1177/088307389901400601. PMID 10385840
- [Result] Cheng J, Xiong Z, Duffney LJ, Wei J, Liu A, Liu S, Chen GJ, Yan Z. Methylphenidate exerts dose-dependent effects on glutamate receptors and behaviors. Biol Psychiatry. 2014 Dec 15;76(12):953-62. doi: 10.1016/j.biopsych.2014.04.003. Epub 2014 Apr 12. PMID 24832867
- [Result] Cherma MD, Josefsson M, Rydberg I, Woxler P, Trygg T, Hollertz O, Gustafsson PA. Methylphenidate for Treating ADHD: A Naturalistic Clinical Study of Methylphenidate Blood Concentrations in Children and Adults With Optimized Dosage. Eur J Drug Metab Pharmacokinet. 2017 Apr;42(2):295-307. doi: 10.1007/s13318-016-0346-1. PMID 27220743
- [Result] Clarke AR, Barry RJ, McCarthy R, Selikowitz M, Croft RJ. EEG differences between good and poor responders to methylphenidate in boys with the inattentive type of attention-deficit/hyperactivity disorder. Clin Neurophysiol. 2002 Aug;113(8):1191-8. doi: 10.1016/s1388-2457(02)00147-5. PMID 12139997
- [Result] Clavenna A, Bonati M. Safety of medicines used for ADHD in children: a review of published prospective clinical trials. Arch Dis Child. 2014 Sep;99(9):866-72. doi: 10.1136/archdischild-2013-304170. Epub 2014 Apr 19. PMID 24748641
- [Result] Coghill DR, Seth S, Pedroso S, Usala T, Currie J, Gagliano A. Effects of methylphenidate on cognitive functions in children and adolescents with attention-deficit/hyperactivity disorder: evidence from a systematic review and a meta-analysis. Biol Psychiatry. 2014 Oct 15;76(8):603-15. doi: 10.1016/j.biopsych.2013.10.005. Epub 2013 Oct 12. PMID 24231201
- [Result] Cortese S, Adamo N, Del Giovane C, Mohr-Jensen C, Hayes AJ, Carucci S, Atkinson LZ, Tessari L, Banaschewski T, Coghill D, Hollis C, Simonoff E, Zuddas A, Barbui C, Purgato M, Steinhausen HC, Shokraneh F, Xia J, Cipriani A. Comparative efficacy and tolerability of medications for attention-deficit hyperactivity disorder in children, adolescents, and adults: a systematic review and network meta-analysis. Lancet Psychiatry. 2018 Sep;5(9):727-738. doi: 10.1016/S2215-0366(18)30269-4. Epub 2018 Aug 7. PMID 30097390
- [Result] Depue BE, Burgess GC, Willcutt EG, Ruzic L, Banich MT. Inhibitory control of memory retrieval and motor processing associated with the right lateral prefrontal cortex: evidence from deficits in individuals with ADHD. Neuropsychologia. 2010 Nov;48(13):3909-17. doi: 10.1016/j.neuropsychologia.2010.09.013. Epub 2010 Sep 21. PMID 20863843
- [Result] Desman C, Petermann F, Hampel P. Deficit in response inhibition in children with attention deficit/hyperactivity disorder (ADHD): impact of motivation? Child Neuropsychol. 2008 Nov;14(6):483-503. doi: 10.1080/09297040701625831. PMID 18982507
- [Result] Dhar M, Been PH, Minderaa RB, Althaus M. Information processing differences and similarities in adults with dyslexia and adults with Attention Deficit Hyperactivity Disorder during a Continuous Performance Test: a study of cortical potentials. Neuropsychologia. 2010 Aug;48(10):3045-56. doi: 10.1016/j.neuropsychologia.2010.06.014. Epub 2010 Jun 17. PMID 20600194
- [Result] Douglas VI, Barr RG, Amin K, O'Neill ME, Britton BG. Dosage effects and individual responsivity to methylphenidate in attention deficit disorder. J Child Psychol Psychiatry. 1988 Jul;29(4):453-75. doi: 10.1111/j.1469-7610.1988.tb00737.x. PMID 3063718
- [Result] Epstein JN, Conners CK, Hervey AS, Tonev ST, Arnold LE, Abikoff HB, Elliott G, Greenhill LL, Hechtman L, Hoagwood K, Hinshaw SP, Hoza B, Jensen PS, March JS, Newcorn JH, Pelham WE, Severe JB, Swanson JM, Wells K, Vitiello B, Wigal T; MTA Cooperative Study Group. Assessing medication effects in the MTA study using neuropsychological outcomes. J Child Psychol Psychiatry. 2006 May;47(5):446-56. doi: 10.1111/j.1469-7610.2005.01469.x. PMID 16671928
- [Result] Epstein JN, Langberg JM, Rosen PJ, Graham A, Narad ME, Antonini TN, Brinkman WB, Froehlich T, Simon JO, Altaye M. Evidence for higher reaction time variability for children with ADHD on a range of cognitive tasks including reward and event rate manipulations. Neuropsychology. 2011 Jul;25(4):427-441. doi: 10.1037/a0022155. PMID 21463041
- [Result] Evans SW, Owens JS, Bunford N. Evidence-based psychosocial treatments for children and adolescents with attention-deficit/hyperactivity disorder. J Clin Child Adolesc Psychol. 2014;43(4):527-51. doi: 10.1080/15374416.2013.850700. Epub 2013 Nov 18. PMID 24245813
- [Result] Faraone SV, Buitelaar J. Comparing the efficacy of stimulants for ADHD in children and adolescents using meta-analysis. Eur Child Adolesc Psychiatry. 2010 Apr;19(4):353-64. doi: 10.1007/s00787-009-0054-3. Epub 2009 Sep 10. PMID 19763664
- [Result] Fayyad J, De Graaf R, Kessler R, Alonso J, Angermeyer M, Demyttenaere K, De Girolamo G, Haro JM, Karam EG, Lara C, Lepine JP, Ormel J, Posada-Villa J, Zaslavsky AM, Jin R. Cross-national prevalence and correlates of adult attention-deficit hyperactivity disorder. Br J Psychiatry. 2007 May;190:402-9. doi: 10.1192/bjp.bp.106.034389. PMID 17470954
- [Result] Fredriksen M, Egeland J, Haavik J, Fasmer OB. Individual Variability in Reaction Time and Prediction of Clinical Response to Methylphenidate in Adult ADHD: A Prospective Open Label Study Using Conners' Continuous Performance Test II. J Atten Disord. 2021 Mar;25(5):657-671. doi: 10.1177/1087054719829822. Epub 2019 Feb 14. PMID 30762452
- [Result] Friehs MA, Frings C. Pimping inhibition: Anodal tDCS enhances stop-signal reaction time. J Exp Psychol Hum Percept Perform. 2018 Dec;44(12):1933-1945. doi: 10.1037/xhp0000579. Epub 2018 Oct 8. PMID 30299126
- [Result] Friehs MA, Frings C. Cathodal tDCS increases stop-signal reaction time. Cogn Affect Behav Neurosci. 2019 Oct;19(5):1129-1142. doi: 10.3758/s13415-019-00740-0. PMID 31313248
- [Result] Fonteneau C, Redoute J, Haesebaert F, Le Bars D, Costes N, Suaud-Chagny MF, Brunelin J. Frontal Transcranial Direct Current Stimulation Induces Dopamine Release in the Ventral Striatum in Human. Cereb Cortex. 2018 Jul 1;28(7):2636-2646. doi: 10.1093/cercor/bhy093. PMID 29688276
- [Result] Fukai M, Bunai T, Hirosawa T, Kikuchi M, Ito S, Minabe Y, Ouchi Y. Endogenous dopamine release under transcranial direct-current stimulation governs enhanced attention: a study with positron emission tomography. Transl Psychiatry. 2019 Mar 15;9(1):115. doi: 10.1038/s41398-019-0443-4. PMID 30877269
- [Result] Gajria K, Lu M, Sikirica V, Greven P, Zhong Y, Qin P, Xie J. Adherence, persistence, and medication discontinuation in patients with attention-deficit/hyperactivity disorder - a systematic literature review. Neuropsychiatr Dis Treat. 2014 Aug 22;10:1543-69. doi: 10.2147/NDT.S65721. eCollection 2014. PMID 25187718
- [Result] Guven A, Altinkaynak M, Dolu N, Demirci E, Ozmen S, Izzetoglu M, Pektas F. Effects of Methylphenidate on Reaction Time in Children with Attention Deficit / Hyperactivity Disorder. Noro Psikiyatr Ars. 2019 Mar;56(1):27-31. doi: 10.29399/npa.22873. Epub 2018 Apr 20. PMID 30911234
- [Result] Hervey AS, Epstein JN, Curry JF, Tonev S, Eugene Arnold L, Keith Conners C, Hinshaw SP, Swanson JM, Hechtman L. Reaction time distribution analysis of neuropsychological performance in an ADHD sample. Child Neuropsychol. 2006 Apr;12(2):125-40. doi: 10.1080/09297040500499081. PMID 16754533
- [Result] Hughes ME, Budd TW, Fulham WR, Lancaster S, Woods W, Rossell SL, Michie PT. Sustained brain activation supporting stop-signal task performance. Eur J Neurosci. 2014 Apr;39(8):1363-9. doi: 10.1111/ejn.12497. Epub 2014 Feb 16. PMID 24528168
- [Result] Huss M, Duhan P, Gandhi P, Chen CW, Spannhuth C, Kumar V. Methylphenidate dose optimization for ADHD treatment: review of safety, efficacy, and clinical necessity. Neuropsychiatr Dis Treat. 2017 Jul 4;13:1741-1751. doi: 10.2147/NDT.S130444. eCollection 2017. PMID 28740389
- [Result] Hood J, Baird G, Rankin PM, Isaacs E. Immediate effects of methylphenidate on cognitive attention skills of children with attention-deficit-hyperactivity disorder. Dev Med Child Neurol. 2005 Jun;47(6):408-14. doi: 10.1017/s0012162205000794. PMID 15934489
- [Result] Inglis SK, Carucci S, Garas P, Hage A, Banaschewski T, Buitelaar JK, Dittmann RW, Falissard B, Hollis C, Kovshoff H, Liddle E, McCarthy S, Nagy P, Neubert A, Rosenthal E, Sonuga-Barke E, Wong I, Zuddas A, Coghill DC; ADDUCE Consortium. Prospective observational study protocol to investigate long-term adverse effects of methylphenidate in children and adolescents with ADHD: the Attention Deficit Hyperactivity Disorder Drugs Use Chronic Effects (ADDUCE) study. BMJ Open. 2016 Apr 26;6(4):e010433. doi: 10.1136/bmjopen-2015-010433. PMID 27118284
- [Result] Iyer MB, Mattu U, Grafman J, Lomarev M, Sato S, Wassermann EM. Safety and cognitive effect of frontal DC brain polarization in healthy individuals. Neurology. 2005 Mar 8;64(5):872-5. doi: 10.1212/01.WNL.0000152986.07469.E9. PMID 15753425
- [Result] Lefaucheur JP, Antal A, Ayache SS, Benninger DH, Brunelin J, Cogiamanian F, Cotelli M, De Ridder D, Ferrucci R, Langguth B, Marangolo P, Mylius V, Nitsche MA, Padberg F, Palm U, Poulet E, Priori A, Rossi S, Schecklmann M, Vanneste S, Ziemann U, Garcia-Larrea L, Paulus W. Evidence-based guidelines on the therapeutic use of transcranial direct current stimulation (tDCS). Clin Neurophysiol. 2017 Jan;128(1):56-92. doi: 10.1016/j.clinph.2016.10.087. Epub 2016 Oct 29. PMID 27866120
- [Result] Lijffijt M, Kenemans JL, Verbaten MN, van Engeland H. A meta-analytic review of stopping performance in attention-deficit/hyperactivity disorder: deficient inhibitory motor control? J Abnorm Psychol. 2005 May;114(2):216-22. doi: 10.1037/0021-843X.114.2.216. PMID 15869352
- [Result] Logan GD, Van Zandt T, Verbruggen F, Wagenmakers EJ. On the ability to inhibit thought and action: general and special theories of an act of control. Psychol Rev. 2014 Jan;121(1):66-95. doi: 10.1037/a0035230. PMID 24490789
- [Result] Lipszyc J, Schachar R. Inhibitory control and psychopathology: a meta-analysis of studies using the stop signal task. J Int Neuropsychol Soc. 2010 Nov;16(6):1064-76. doi: 10.1017/S1355617710000895. Epub 2010 Aug 19. PMID 20719043
- [Result] Logan GD, Cowan WB, Davis KA. On the ability to inhibit simple and choice reaction time responses: a model and a method. J Exp Psychol Hum Percept Perform. 1984 Apr;10(2):276-91. doi: 10.1037//0096-1523.10.2.276. PMID 6232345
- [Result] MacDonald SW, Nyberg L, Backman L. Intra-individual variability in behavior: links to brain structure, neurotransmission and neuronal activity. Trends Neurosci. 2006 Aug;29(8):474-80. doi: 10.1016/j.tins.2006.06.011. Epub 2006 Jul 3. PMID 16820224
- [Result] Mannuzza S, Klein RG, Bessler A, Malloy P, LaPadula M. Adult outcome of hyperactive boys. Educational achievement, occupational rank, and psychiatric status. Arch Gen Psychiatry. 1993 Jul;50(7):565-76. doi: 10.1001/archpsyc.1993.01820190067007. PMID 8317950
- [Result] Marcos E, Pani P, Brunamonti E, Deco G, Ferraina S, Verschure P. Neural variability in premotor cortex is modulated by trial history and predicts behavioral performance. Neuron. 2013 Apr 24;78(2):249-55. doi: 10.1016/j.neuron.2013.02.006. PMID 23622062
- [Result] McLaren ME, Nissim NR, Woods AJ. The effects of medication use in transcranial direct current stimulation: A brief review. Brain Stimul. 2018 Jan-Feb;11(1):52-58. doi: 10.1016/j.brs.2017.10.006. Epub 2017 Oct 12. PMID 29066167
- [Result] Menghini D, Armando M, Calcagni M, Napolitano C, Pasqualetti P, Sergeant JA, Pani P, Vicari S. The influence of Generalized Anxiety Disorder on Executive Functions in children with ADHD. Eur Arch Psychiatry Clin Neurosci. 2018 Jun;268(4):349-357. doi: 10.1007/s00406-017-0831-9. Epub 2017 Aug 1. PMID 28766128
- [Result] Molina BSG, Hinshaw SP, Swanson JM, Arnold LE, Vitiello B, Jensen PS, Epstein JN, Hoza B, Hechtman L, Abikoff HB, Elliott GR, Greenhill LL, Newcorn JH, Wells KC, Wigal T, Gibbons RD, Hur K, Houck PR; MTA Cooperative Group. The MTA at 8 years: prospective follow-up of children treated for combined-type ADHD in a multisite study. J Am Acad Child Adolesc Psychiatry. 2009 May;48(5):484-500. doi: 10.1097/CHI.0b013e31819c23d0. PMID 19318991
- [Result] Monte-Silva K, Kuo MF, Hessenthaler S, Fresnoza S, Liebetanz D, Paulus W, Nitsche MA. Induction of late LTP-like plasticity in the human motor cortex by repeated non-invasive brain stimulation. Brain Stimul. 2013 May;6(3):424-32. doi: 10.1016/j.brs.2012.04.011. Epub 2012 Jun 2. PMID 22695026
- [Result] Nigg JT, Casey BJ. An integrative theory of attention-deficit/ hyperactivity disorder based on the cognitive and affective neurosciences. Dev Psychopathol. 2005 Summer;17(3):785-806. doi: 10.1017/S0954579405050376. PMID 16262992
- [Result] Nitsche MA, Paulus W. Excitability changes induced in the human motor cortex by weak transcranial direct current stimulation. J Physiol. 2000 Sep 15;527 Pt 3(Pt 3):633-9. doi: 10.1111/j.1469-7793.2000.t01-1-00633.x. PMID 10990547
- [Result] Nitsche MA, Cohen LG, Wassermann EM, Priori A, Lang N, Antal A, Paulus W, Hummel F, Boggio PS, Fregni F, Pascual-Leone A. Transcranial direct current stimulation: State of the art 2008. Brain Stimul. 2008 Jul;1(3):206-23. doi: 10.1016/j.brs.2008.06.004. Epub 2008 Jul 1. PMID 20633386
- [Result] Nitsche MA, Boggio PS, Fregni F, Pascual-Leone A. Treatment of depression with transcranial direct current stimulation (tDCS): a review. Exp Neurol. 2009 Sep;219(1):14-9. doi: 10.1016/j.expneurol.2009.03.038. Epub 2009 Apr 5. PMID 19348793
- [Result] Oosterlaan J, Logan GD, Sergeant JA. Response inhibition in AD/HD, CD, comorbid AD/HD + CD, anxious, and control children: a meta-analysis of studies with the stop task. J Child Psychol Psychiatry. 1998 Mar;39(3):411-25. PMID 9670096
- [Result] Johnson KA, Kelly SP, Bellgrove MA, Barry E, Cox M, Gill M, Robertson IH. Response variability in attention deficit hyperactivity disorder: evidence for neuropsychological heterogeneity. Neuropsychologia. 2007 Mar 2;45(4):630-8. doi: 10.1016/j.neuropsychologia.2006.03.034. Epub 2006 Dec 8. PMID 17157885
- [Result] Kim S, Stephenson MC, Morris PG, Jackson SR. tDCS-induced alterations in GABA concentration within primary motor cortex predict motor learning and motor memory: a 7 T magnetic resonance spectroscopy study. Neuroimage. 2014 Oct 1;99:237-43. doi: 10.1016/j.neuroimage.2014.05.070. Epub 2014 Jun 3. PMID 24904994
- [Result] KIRCHNER WK. Age differences in short-term retention of rapidly changing information. J Exp Psychol. 1958 Apr;55(4):352-8. doi: 10.1037/h0043688. No abstract available. PMID 13539317
- [Result] Klein RM, Castel AD, Pratt J. The effects of memory load on the time course of inhibition of return. Psychon Bull Rev. 2006 Apr;13(2):294-9. doi: 10.3758/bf03193846. PMID 16892997
- [Result] Klorman R, Brumaghim JT, Fitzpatrick PA, Borgstedt AD. Methylphenidate reduces abnormalities of stimulus classification in adolescents with attention deficit disorder. J Abnorm Psychol. 1992 Feb;101(1):130-8. doi: 10.1037//0021-843x.101.1.130. PMID 1537959
- [Result] Klorman R, Brumaghim JT, Salzman LF, Strauss J, Borgstedt AD, McBride MC, Loeb S. Effects of methylphenidate on processing negativities in patients with attention-deficit hyperactivity disorder. Psychophysiology. 1990 May;27(3):328-37. doi: 10.1111/j.1469-8986.1990.tb00391.x. PMID 2236435
- [Result] Klotz JM, Johnson MD, Wu SW, Isaacs KM, Gilbert DL. Relationship between reaction time variability and motor skill development in ADHD. Child Neuropsychol. 2012;18(6):576-85. doi: 10.1080/09297049.2011.625356. Epub 2011 Nov 24. PMID 22111593
- [Result] Kofler MJ, Rapport MD, Sarver DE, Raiker JS, Orban SA, Friedman LM, Kolomeyer EG. Reaction time variability in ADHD: a meta-analytic review of 319 studies. Clin Psychol Rev. 2013 Aug;33(6):795-811. doi: 10.1016/j.cpr.2013.06.001. Epub 2013 Jun 13. PMID 23872284
- [Result] Konrad K, Gunther T, Heinzel-Gutenbrunner M, Herpertz-Dahlmann B. Clinical evaluation of subjective and objective changes in motor activity and attention in children with attention-deficit/hyperactivity disorder in a double-blind methylphenidate trial. J Child Adolesc Psychopharmacol. 2005 Apr;15(2):180-90. doi: 10.1089/cap.2005.15.180. PMID 15910203
- [Result] Krishnan C, Santos L, Peterson MD, Ehinger M. Safety of noninvasive brain stimulation in children and adolescents. Brain Stimul. 2015 Jan-Feb;8(1):76-87. doi: 10.1016/j.brs.2014.10.012. Epub 2014 Oct 28. PMID 25499471
- [Result] Kuntsi J, Klein C. Intraindividual variability in ADHD and its implications for research of causal links. Curr Top Behav Neurosci. 2012;9:67-91. doi: 10.1007/7854_2011_145. PMID 21769722
- [Result] Kuo MF, Paulus W, Nitsche MA. Boosting focally-induced brain plasticity by dopamine. Cereb Cortex. 2008 Mar;18(3):648-51. doi: 10.1093/cercor/bhm098. Epub 2007 Jun 24. PMID 17591596
- [Result] Kuo MF, Paulus W, Nitsche MA. Therapeutic effects of non-invasive brain stimulation with direct currents (tDCS) in neuropsychiatric diseases. Neuroimage. 2014 Jan 15;85 Pt 3:948-60. doi: 10.1016/j.neuroimage.2013.05.117. Epub 2013 Jun 4. PMID 23747962
- [Result] Palm U, Keeser D, Schiller C, Fintescu Z, Nitsche M, Reisinger E, Padberg F. Skin lesions after treatment with transcranial direct current stimulation (tDCS). Brain Stimul. 2008 Oct;1(4):386-7. doi: 10.1016/j.brs.2008.04.003. Epub 2008 Jun 20. No abstract available. PMID 20633396
- [Result] Pani P, Menghini D, Napolitano C, Calcagni M, Armando M, Sergeant JA, Vicari S. Proactive and reactive control of movement are differently affected in Attention Deficit Hyperactivity Disorder children. Res Dev Disabil. 2013 Oct;34(10):3104-11. doi: 10.1016/j.ridd.2013.06.032. Epub 2013 Jul 22. PMID 23886755
- [Result] Pauls AM, O'Daly OG, Rubia K, Riedel WJ, Williams SC, Mehta MA. Methylphenidate effects on prefrontal functioning during attentional-capture and response inhibition. Biol Psychiatry. 2012 Jul 15;72(2):142-9. doi: 10.1016/j.biopsych.2012.03.028. Epub 2012 May 1. PMID 22552046
- [Result] Polanczyk GV, Willcutt EG, Salum GA, Kieling C, Rohde LA. ADHD prevalence estimates across three decades: an updated systematic review and meta-regression analysis. Int J Epidemiol. 2014 Apr;43(2):434-42. doi: 10.1093/ije/dyt261. Epub 2014 Jan 24. PMID 24464188
- [Result] Poreisz C, Boros K, Antal A, Paulus W. Safety aspects of transcranial direct current stimulation concerning healthy subjects and patients. Brain Res Bull. 2007 May 30;72(4-6):208-14. doi: 10.1016/j.brainresbull.2007.01.004. Epub 2007 Jan 24. PMID 17452283
- [Result] Rapport MD, DuPaul GJ, Kelly KL. Attention deficit hyperactivity disorder and methylphenidate: the relationship between gross body weight and drug response in children. Psychopharmacol Bull. 1989;25(2):285-90. No abstract available. PMID 2602521
- [Result] Rosch KS, Fosco WD, Pelham WE Jr, Waxmonsky JG, Bubnik MG, Hawk LW Jr. Reinforcement and Stimulant Medication Ameliorate Deficient Response Inhibition in Children with Attention-Deficit/Hyperactivity Disorder. J Abnorm Child Psychol. 2016 Feb;44(2):309-21. doi: 10.1007/s10802-015-0031-x. PMID 25985978
- [Result] Rubia K, Halari R, Cubillo A, Mohammad AM, Brammer M, Taylor E. Methylphenidate normalises activation and functional connectivity deficits in attention and motivation networks in medication-naive children with ADHD during a rewarded continuous performance task. Neuropharmacology. 2009 Dec;57(7-8):640-52. doi: 10.1016/j.neuropharm.2009.08.013. Epub 2009 Aug 26. PMID 19715709
- [Result] Russell VA, Oades RD, Tannock R, Killeen PR, Auerbach JG, Johansen EB, Sagvolden T. Response variability in Attention-Deficit/Hyperactivity Disorder: a neuronal and glial energetics hypothesis. Behav Brain Funct. 2006 Aug 23;2:30. doi: 10.1186/1744-9081-2-30. PMID 16925830
- [Result] Simon V, Czobor P, Balint S, Meszaros A, Bitter I. Prevalence and correlates of adult attention-deficit hyperactivity disorder: meta-analysis. Br J Psychiatry. 2009 Mar;194(3):204-11. doi: 10.1192/bjp.bp.107.048827. PMID 19252145
- [Result] Salehinejad MA, Wischnewski M, Nejati V, Vicario CM, Nitsche MA. Transcranial direct current stimulation in attention-deficit hyperactivity disorder: A meta-analysis of neuropsychological deficits. PLoS One. 2019 Apr 12;14(4):e0215095. doi: 10.1371/journal.pone.0215095. eCollection 2019. PMID 30978259
- [Result] Schachar R, Ickowicz A, Crosbie J, Donnelly GA, Reiz JL, Miceli PC, Harsanyi Z, Darke AC. Cognitive and behavioral effects of multilayer-release methylphenidate in the treatment of children with attention-deficit/hyperactivity disorder. J Child Adolesc Psychopharmacol. 2008 Feb;18(1):11-24. doi: 10.1089/cap.2007.0039. PMID 18294084
- [Result] Soltaninejad Z, Nejati V, Ekhtiari H. Effect of Anodal and Cathodal Transcranial Direct Current Stimulation on DLPFC on Modulation of Inhibitory Control in ADHD. J Atten Disord. 2019 Feb;23(4):325-332. doi: 10.1177/1087054715618792. Epub 2015 Dec 20. PMID 26689935
- [Result] Soff C, Sotnikova A, Christiansen H, Becker K, Siniatchkin M. Transcranial direct current stimulation improves clinical symptoms in adolescents with attention deficit hyperactivity disorder. J Neural Transm (Vienna). 2017 Jan;124(1):133-144. doi: 10.1007/s00702-016-1646-y. Epub 2016 Nov 16. PMID 27853926
- [Result] Solanto MV. Behavioral effects of low-dose methylphenidate in childhood attention deficit disorder: implications for a mechanism of stimulant drug action. J Am Acad Child Psychiatry. 1986 Jan;25(1):96-101. doi: 10.1016/s0002-7138(09)60604-x. No abstract available. PMID 3950273
- [Result] Solanto MV. Dopamine dysfunction in AD/HD: integrating clinical and basic neuroscience research. Behav Brain Res. 2002 Mar 10;130(1-2):65-71. doi: 10.1016/s0166-4328(01)00431-4. PMID 11864719
- [Result] Sonuga-Barke EJ, Sergeant JA, Nigg J, Willcutt E. Executive dysfunction and delay aversion in attention deficit hyperactivity disorder: nosologic and diagnostic implications. Child Adolesc Psychiatr Clin N Am. 2008 Apr;17(2):367-84, ix. doi: 10.1016/j.chc.2007.11.008. PMID 18295151
- [Result] Spencer SV, Hawk LW Jr, Richards JB, Shiels K, Pelham WE Jr, Waxmonsky JG. Stimulant treatment reduces lapses in attention among children with ADHD: the effects of methylphenidate on intra-individual response time distributions. J Abnorm Child Psychol. 2009 Aug;37(6):805-16. doi: 10.1007/s10802-009-9316-2. PMID 19291387
- [Result] Stein MA, Sarampote CS, Waldman ID, Robb AS, Conlon C, Pearl PL, Black DO, Seymour KE, Newcorn JH. A dose-response study of OROS methylphenidate in children with attention-deficit/hyperactivity disorder. Pediatrics. 2003 Nov;112(5):e404. doi: 10.1542/peds.112.5.e404. PMID 14595084
- [Result] Tamm L, Narad ME, Antonini TN, O'Brien KM, Hawk LW Jr, Epstein JN. Reaction time variability in ADHD: a review. Neurotherapeutics. 2012 Jul;9(3):500-8. doi: 10.1007/s13311-012-0138-5. PMID 22930417
- [Result] Tannock R, Ickowicz A, Schachar R. Differential effects of methylphenidate on working memory in ADHD children with and without comorbid anxiety. J Am Acad Child Adolesc Psychiatry. 1995 Jul;34(7):886-96. doi: 10.1097/00004583-199507000-00012. PMID 7649959
- [Result] Vaurio RG, Simmonds DJ, Mostofsky SH. Increased intra-individual reaction time variability in attention-deficit/hyperactivity disorder across response inhibition tasks with different cognitive demands. Neuropsychologia. 2009 Oct;47(12):2389-96. doi: 10.1016/j.neuropsychologia.2009.01.022. Epub 2009 Jan 22. PMID 19552927
- [Result] Volkow ND, Wang GJ, Fowler JS, Gatley SJ, Logan J, Ding YS, Hitzemann R, Pappas N. Dopamine transporter occupancies in the human brain induced by therapeutic doses of oral methylphenidate. Am J Psychiatry. 1998 Oct;155(10):1325-31. doi: 10.1176/ajp.155.10.1325. PMID 9766762
- [Result] Wigal SB, Nordbrock E, Adjei AL, Childress A, Kupper RJ, Greenhill L. Efficacy of Methylphenidate Hydrochloride Extended-Release Capsules (Aptensio XR) in Children and Adolescents with Attention-Deficit/Hyperactivity Disorder: A Phase III, Randomized, Double-Blind Study. CNS Drugs. 2015 Apr;29(4):331-40. doi: 10.1007/s40263-015-0241-3. PMID 25877989
- [Result] Willcutt EG, Doyle AE, Nigg JT, Faraone SV, Pennington BF. Validity of the executive function theory of attention-deficit/hyperactivity disorder: a meta-analytic review. Biol Psychiatry. 2005 Jun 1;57(11):1336-46. doi: 10.1016/j.biopsych.2005.02.006. PMID 15950006
- [Result] Williams BR, Ponesse JS, Schachar RJ, Logan GD, Tannock R. Development of inhibitory control across the life span. Dev Psychol. 1999 Jan;35(1):205-13. doi: 10.1037//0012-1649.35.1.205. PMID 9923475
- [Result] Costanzo F, Menghini D, Casula L, Amendola A, Mazzone L, Valeri G, Vicari S. Transcranial Direct Current Stimulation Treatment in an Adolescent with Autism and Drug-Resistant Catatonia. Brain Stimul. 2015 Nov-Dec;8(6):1233-5. doi: 10.1016/j.brs.2015.08.009. Epub 2015 Aug 24. No abstract available. PMID 26590479
- [Result] Costanzo F, Varuzza C, Rossi S, Sdoia S, Varvara P, Oliveri M, Koch G, Vicari S, Menghini D. Reading changes in children and adolescents with dyslexia after transcranial direct current stimulation. Neuroreport. 2016 Mar 23;27(5):295-300. doi: 10.1097/WNR.0000000000000536. PMID 26848997
- [Result] Costanzo F, Varuzza C, Rossi S, Sdoia S, Varvara P, Oliveri M, Giacomo K, Vicari S, Menghini D. Evidence for reading improvement following tDCS treatment in children and adolescents with Dyslexia. Restor Neurol Neurosci. 2016;34(2):215-26. doi: 10.3233/RNN-150561. PMID 26890096
- [Result] Costanzo F, Rossi S, Varuzza C, Varvara P, Vicari S, Menghini D. Long-lasting improvement following tDCS treatment combined with a training for reading in children and adolescents with dyslexia. Neuropsychologia. 2019 Jul;130:38-43. doi: 10.1016/j.neuropsychologia.2018.03.016. Epub 2018 Mar 14. PMID 29550525
- [Result] Costanzo F, Menghini D, Maritato A, Castiglioni MC, Mereu A, Varuzza C, Zanna V, Vicari S. New Treatment Perspectives in Adolescents With Anorexia Nervosa: The Efficacy of Non-invasive Brain-Directed Treatment. Front Behav Neurosci. 2018 Jul 20;12:133. doi: 10.3389/fnbeh.2018.00133. eCollection 2018. PMID 30083095
- [Result] Lazzaro G, Bertoni S, Menghini D, Costanzo F, Franceschini S, Varuzza C, Ronconi L, Battisti A, Gori S, Facoetti A, Vicari S. Beyond Reading Modulation: Temporo-Parietal tDCS Alters Visuo-Spatial Attention and Motion Perception in Dyslexia. Brain Sci. 2021 Feb 19;11(2):263. doi: 10.3390/brainsci11020263. PMID 33669651
- [Result] Lazzaro G, Costanzo F, Varuzza C, Rossi S, Vicari S, Menghini D. Effects of a short, intensive, multi-session tDCS treatment in developmental dyslexia: Preliminary results of a sham-controlled randomized clinical trial. Prog Brain Res. 2021;264:191-210. doi: 10.1016/bs.pbr.2021.01.015. PMID 34167656